CLINICAL TRIAL: NCT03163485
Title: Prospective, Open Label, Multi-centre, Controlled Phase 2a Clinical Trial to Investigate the Safety and Diagnostic Performance of the Multifunctional Hybrid Device Combining a Micro-dialysis Probe With an Intra-cortical Depth Electrode (DIALYTRODE) for Short Time Continuous Multimodal Neuro-monitoring of NICU Patients With Severe Brain Injury and Suspected Status Epilepticus in Surface EEG
Brief Title: Hybrid Device DIALYTRODE for Multimodal Neuro-monitoring of Patients With Brain Injury and Status Epilepticus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Application to CA withdrawn due to technical reasons of the manufacturer
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: European Commission (Other); University of Aarhus (Other); Royal College of Surgeons, Ireland (Other); Philipps University Marburg (Other); Dixi Medical (Unknown); ARTTIC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UKER-EPIMI-RNA-C
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy; Brain Injuries
Keywords: epilepsy; multimodal neuromonitoring; depth EEG; microdialysis; brain injury; brain tissue at risk; NCSE; short time monitoring; neurologic ICU
MeSH Terms: conditions — Epilepsy; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialytrode (Experimental): Multimodal neuro-monitoring by dialytrode (investigational medical device)
  Interventions: Device: Dialytrode
- Standard treatment (Other): Either EVD and/or micro-dialysis according to standard treatment
  Interventions: Device: Standard treatment

INTERVENTIONS:
Device: Dialytrode — Multimodal neuromonitoring by intracerebral depth EEG recording combined with microdialysis for the sampling of cerebrospinal fluid during EEG recording
  Arms: Dialytrode
Device: Standard treatment — Monitoring of intracranial pressure by EVD and/or multimodal neuromonitoring by microdialysis for sampling of cerebrospinal fluid
  Other Names: EVD and/or microdialysis catheter alone
  Arms: Standard treatment

SUMMARY:
This clinical trial evaluates the safety and diagnostic performance of a newly developed combined catheter that will be implanted into the brain of patients with severe brain injury for short time (up to 28 days) monitoring of the electric activity and the metabolism of brain tissue at risk. Ten patients will be monitored with the new device and seven patients will be monitored by intracerebral probes according to standard treatment.

DETAILED DESCRIPTION:
Early detection of nonconvulsive status epilepticus (NCSE) in patients treated in neurological intensive care unit (NICU) is essential, as delayed treatment can aggravate their clinical situation and worsen the outcome. In this study in intensive care patients with severe brain injury due to malignant middle cerebral artery (MCA) infarction, subarachnoidal hemorrhage (SAH) or intracerebral hemorrhage (ICH) with suspected status epilepticus in the surface EEG the hybrid catheter Dialytrode will be implanted in the cortical brain tissue by neurosurgeons for short time continuous bedside multimodal neuro-monitoring. Dialytrode combines a microdialysis catheter and depth EEG probe. Ten subjects will be monitored by Dialytrode and an additional (intracranial pressure (ICP) probe. Subjects with an clinical indication of an external ventricular drain (EVD) or cerebral microdialysis alone serve as control. The monitoring period with the device is limited to the microdialysis phase with a maximum of 28 days. Subjects will be followed up for 7 days after end of intracerebral monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical condition requiring treatment in NICU
2. MCA OR Subarachnoidal haemorrhage (SAH) OR Intracerebral haemorrhage (ICH)
3. Given indication of EVD with or without multimodal monitoring by micro-dialysis OR Given indication of multimodal monitoring by micro-dialysis and continuous depth EEG-monitoring due to (a) suspected SE in surface EEG (e.g. rhythmic pattern) or (b) refractory status epilepticus (RSE) in surface EEG or (c) an unclear situation of not waking up even though sedation is reduced OR Suspected SE without acute brain injury

Exclusion Criteria (main criteria):

* Subject receiving anticoagulants in therapeutic dose
* Bleeding disorder
* Known contraindications for EEG depth electrodes or microdialysis probes
* Presence of an infectious lesion of skin (limited to the scalp)
* Presence of general contraindications for any surgical intervention
* Sepsis or acute severe bacterial infection
* Fragile bones of the skull
* Severe organ failure or medical conditions displaying a contraindication for participating
* Pregnant or nursing woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-06-25 (Estimated); Study Completion 2020-07-25 (Estimated)

PRIMARY OUTCOMES:
Number of adverse device effects (ADE) and serious adverse device effects (SADE) | Up to day 7±2 after removal of IMD or the single control devices respectively
  Number of adverse device effects (ADE) and serious adverse device effects (SADE) from Baseline (day 1) to day 7+/-2 after removal of the investigational medical device (IMD) or the control devices respectively) in the intervention group compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Hajo Hamer, MD PhD, Principal Investigator — Universitätsklinikum Erlangen Neurologische Klinik
Locations (2):
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt Epilepsiezentrum Rhein-Main, Frankfurt am Main

IPD SHARING:
Plan to Share IPD: Undecided